CLINICAL TRIAL: NCT06607575
Title: The Effect of Warming and Vibration Applications on Pain During Heel Blood Collection in Newborns
Brief Title: The Effect of Warming and Vibration Applications on Pain in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2023-10/403
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Pain
Keywords: Newborn; pain; vibration; warming; heel blood collection; infant
MeSH Terms: conditions — Pain | interventions — Control Groups; Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Other): Newborns who will be subjected to routine practices during heel blood collection procedure and who will not be subjected to warming and vibration will constitute the control group.
  Interventions: Other: Control group
- Experimental group (warming) (Experimental): Newborns who will be subjected to warming application during the heel blood collection procedure will constitute the 1st experimental group.
  Interventions: Other: Warming
- Experimental group (vibration) (Experimental): Newborns who will be subjected to vibration during the heel blood collection procedure will constitute the 2nd experimental group.
  Interventions: Other: Vibration
- Experimental group (warming and vibration) (Experimental): Newborns who will be subjected to both warming and vibration during the heel blood collection procedure will constitute the 3rd experimental group.
  Interventions: Other: Warming and vibration

INTERVENTIONS:
Other: Control group — 1. The procedure for heel blood collection will be performed.
  2. Pain assessment will be performed with the N-PASS scale during and after the procedure.
  Arms: Control group
Other: Warming — 1. The cotton sock will be warmed under the heater for 3 minutes. The sock will be put on the newborn and taken off after 3 minutes.
  2. The procedure for heel blood collection will be performed.
  3. Pain assessment will be performed with the N-PASS scale during and after the procedure.
  Arms: Experimental group (warming)
Other: Vibration — 1. A rechargeable toothbrush will be prepared for the newborn to whom vibration will be applied. The vibration process will be applied to the midline of the gastrocnemius muscle for 3 minutes.
  2. The procedure for heel blood collection will be performed.
  3. Pain assessment will be performed with the N-PASS scale during and after the procedure.
  Arms: Experimental group (vibration)
Other: Warming and vibration — 1. After the socks are warmed, they will be put on the newborn's feet and both warming and vibration will be applied for 3 minutes.
  2. The procedure for heel blood collection will be performed.
  3. Pain assessment will be performed with the N-PASS scale during and after the procedure.
  Arms: Experimental group (warming and vibration)

SUMMARY:
This study aimed to determine the effects of warming and vibration applications on pain during heel blood collection in newborns.

H1: Warming application has a positive effect on pain during heel blood collection in newborns.

H2: Vibration application has a positive effect on pain during heel blood collection in newborns.

H3: The combined application of warming and vibration during heel blood collection in newborns has a positive effect on pain.

DETAILED DESCRIPTION:
Heel blood collection is frequently used for neonatal metabolic screening and analysis of bilirubin, glucose and other biochemical/hematologic parameters. This process is both painful and stressful for the newborn. Pain experience in the neonatal period can cause intense stress in the infant and cause physiopathological changes such as respiratory irregularity, impaired thermoregulation, changes in heart rhythm, changes in oxygen saturation and blood pressure. Therefore, it is recommended to use evidence-based non-pharmacological methods to reduce the pain experiences of newborns and to minimize the short and long-term negative effects of pain.

Based on this rationale, this study was planned to evaluate the effect of non-pharmacologic methods on pain and procedure time together.

ELIGIBILITY:
Inclusion Criteria:

* Newborns at 38 weeks of gestation and above
* Healthy newborns

Exclusion Criteria:

* Newborns with any lower extremity anomalies
* Newborns with congenital diseases

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Change in level of pain | Immediately before the prosedure, during the procedure, immediately after the procedure. The change in these time period will be measured.
  The level of pain will be measured using the N-PASS: Neonatal Pain/Agitation, Sedation Scale. The scale was developed by Hummel, Lawlor-Klean and Weiss in 2010, its Turkish validity and reliability were made by Açıkgöz et al. in 2017. N-PASS consists of two sections: sedation and pain assessment. Total pain score varies between 0 and +11 and total sedation score varies between 0 and +10. A high score indicates severe pain. The aim is to keep the score at 3 and below. If it is above 3 points, sedation requirements are evaluated. The average time spent to administer the scale is 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Keskin Nurse, Principal Investigator — Acibadem University
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University, Istanbul, Ata
  - Acıbadem University, Istanbul, Ataşehir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avan Antepli N, Bilsin Kocamaz E, Gungormus Z. The Effect of Vibration on Pain During Heel Lance Procedures in Newborns: A Randomized Controlled Trial. Adv Neonatal Care. 2022 Apr 1;22(2):E43-E47. doi: 10.1097/ANC.0000000000000918. PMID 34334677
- [Background] Shepherd AJ, Glenesk A, Niven CA, Mackenzie J. A Scottish study of heel-prick blood sampling in newborn babies. Midwifery. 2006 Jun;22(2):158-68. doi: 10.1016/j.midw.2005.07.002. Epub 2005 Dec 28. PMID 16386341
- [Background] Ray R, Godwin Y, Shepherd A. Convective burn from use of hairdryer for heel warming prior to the heel prick test - a case report. BMC Pediatr. 2011 May 10;11:30. doi: 10.1186/1471-2431-11-30. PMID 21569274
- [Background] Napiorkowska-Orkisz M, Gutysz-Wojnicka A, Tanajewska M, Sadowska-Krawczenko I. Evaluation of Methods to Minimize Pain in Newborns during Capillary Blood Sampling for Screening: A Randomized Clinical Trial. Int J Environ Res Public Health. 2022 Jan 13;19(2):870. doi: 10.3390/ijerph19020870. PMID 35055694
- [Background] Hassan Z, Shah M. Scald injury from the Guthrie test: should the heel be warmed? Arch Dis Child Fetal Neonatal Ed. 2005 Nov;90(6):F533-4. doi: 10.1136/adc.2005.072678. PMID 16244215